CLINICAL TRIAL: NCT04605224
Title: Effectiveness of a Culinary Class on Food Literacy and Eating Behaviours of Francophone High School Students
Status: Completed | Type: Observational
Sponsor: Universite de Moncton (Other)
Responsible Party: Principal Investigator, Stephanie Ward, Adjunct Professor, Universite de Moncton
Other Study IDs: 1920-002
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Eating Behavior; Fruit and Vegetable Intake
Keywords: School; Cooking class; Culinary class; Food literacy; Cooking skills; Food skills
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Culinary class (intervention group): The culinary class is 55-70 minutes in duration and is offered daily, Monday to Friday, over an 18-week semester (September 2019 to January 2020).
  Interventions: Behavioral: Culinary class
- Social studies class (control group): The social studies class is 55-70 minutes in duration and is offered daily, Monday to Friday, over an 18-week semester (September 2019 to January 2020).

INTERVENTIONS:
Behavioral: Culinary class — This hands-on, optional course teaches students how to measure and weigh ingredients, read and follow recipes, apply various food preparation, cooking and assembly techniques, as well as prepare meals, as per the provincial curriculum
  Other Names: Cuisine professionnelle
  Groups: Culinary class (intervention group)

SUMMARY:
As the frequency of meals taken outside the home increases, children and youth have less opportunities to develop their food and cooking skills. Consequently, poor food literacy can increase dependence on highly processed foods which generally contain high amounts of calories, fat, sugar and sodium. Past studies have shown positive impacts of culinary-based interventions on adolescents' nutrition knowledge, attitudes, eating behaviours and cooking skills. However, most of these interventions were led outside of the school context, which limits their reach. Since adolescents spend most of their waking hours in school, providing culinary classes in school may be an effective way of promoting adolescents' food literacy. Therefore, the aim of this quasi-experimental study was to assess the effectiveness of an optional culinary class on high school students' food literacy and eating behaviours. Specifically, data were collected among students from five francophone high schools who were enrolled in a culinary class. These students were compared to those who were enrolled in a social studies class. Both classes were 55-70 minutes in duration and were provided five times per week over a full 18-week semester. Data on students' food literacy and eating behaviours were collected via questionnaires during the first and last week of the semester.

DETAILED DESCRIPTION:
This study used a quasi-experimental design. Students from five francophone high schools in the province of New Brunswick, Canada, who were enrolled in an optional culinary class were compared to students from those same schools who were enrolled in a social studies class. The culinary class is a hands-on course which teaches students how to measure and weigh ingredients, read and follow recipes, apply various food preparation, cooking and assembly techniques, as well as prepare meals. In contrast, the social studies class is a mandatory theory-based course which teaches students how to maintain positive relationships, how to become a productive member of society and how to make responsible and informed choices related to their health. Both classes are 55-70 minutes in duration and are provided daily over an 18-week semester.

A questionnaire was developed based on two previously validated food literacy questionnaires and assessed food and cooking skills, as well as eating behaviours. This pen and paper questionnaire was completed by students in both the culinary class and the social studies class during the first and last week of the semester (September 2019 and January 2020). Multilevel regressions will be used to assess the effectiveness of the culinary class on students' food literacy and eating behaviours as compared to the social studies class.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in either the culinary class or social studies class in the fall semester of 2019

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants are students enrolled in the Culinary class or Social Studies class in the fall of 2019, in the 5 recruited francophone high schools in the province of New Brunswick, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cooking skills at the end of the school semester | Baseline and Week 18
  The validated 14-item cooking skills question assesses how good students feel they are at performing each cooking skill on a scale from 1 (very poor) to 7 (very good) with the option "Never/rarely do it" (0) given as an option. Change is measured by the difference between the total score (0 to 98) obtained at the end of the semester (18 weeks) minus the total score obtained at baseline.
Change from baseline in food skills at the end of the school semester | Baseline and Week 18
  The validated 12-item food skills question assesses how good students feel they are at performing each food skill on a scale from 1 (very poor) to 7 (very good) with the option "Never/rarely do it" (0) given as an option. Change is measured by the difference between the total score (0 to 84) obtained at the end of the semester (18 weeks) minus the total score obtained at baseline.
Change from baseline in eating behaviours at the end of the school semester | Baseline and Week 18
  Eating behaviours were measured using two separate questions. The first question, based on the NB Student Wellness Survey, assessed how often students consumed breakfast in the previous week (0 pt = never to 7 pt = 7 times).
  The second question was based on a previously validated questionnaire. This question assessed how often students did 6 different eating related behaviours. Response options ranged from "never or rarely" (0 pt) to "every day" (3 pts), for a maximum total score of 18 points.
  These two questions were combined to provide a total score ranging from 0 to 25 points. Change is measured by the difference between the total score (0 to 25) obtained at the end of the semester (18 weeks) minus the total score obtained at baseline.
Change from baseline in fruit and vegetable intake at the end of the school semester | Baseline and Week 18
  Intake was measured using 7 items of a previously validated questionnaire. One question assessed how many servings of vegetables and how many servings of fruit they usually eat each day. Response options ranged from "I don't eat vegetables/fruit" (0 pt) to "more than 5 servings per day" (5 pts). Another question assessed whether students had eaten or were planning on eating various types of foods at breakfast, lunch or snack that day. One point was given every time a vegetable or fruit product was checked, for a maximum of 9 points. A third question assessed whether they had consumed the listed fruit or vegetable the previous day. Scores ranged from 0 to 4 points.
  The sum of these questions provided a total possible score of 25 points. Change is measured by the difference between the total score (0 to 25) obtained at the end of the semester (18 weeks) minus the total score obtained at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Ward, PhD, RD, Principal Investigator — Universite de Moncton
Locations (1):
- Universite de Moncton, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be made available to researchers upon reasonable request made to the principal investigator.

REFERENCES:
- [Background] Lavelle F, McGowan L, Hollywood L, Surgenor D, McCloat A, Mooney E, Caraher M, Raats M, Dean M. The development and validation of measures to assess cooking skills and food skills. Int J Behav Nutr Phys Act. 2017 Sep 2;14(1):118. doi: 10.1186/s12966-017-0575-y. PMID 28865452
- [Background] Wilson AM, Magarey AM, Mastersson N. Reliability and relative validity of a child nutrition questionnaire to simultaneously assess dietary patterns associated with positive energy balance and food behaviours, attitudes, knowledge and environments associated with healthy eating. Int J Behav Nutr Phys Act. 2008 Jan 29;5:5. doi: 10.1186/1479-5868-5-5. PMID 18226268